CLINICAL TRIAL: NCT05196633
Title: Effectiveness of Radial Extracorporeal Shock Wave Therapy and Visual Feedback Balance Training on Lower Limb Post-Stroke Spasticity, Trunk Performance and Balance: A Randomized Controlled Trial
Brief Title: Radial Extracorporeal Shock Wave Therapy and Visual Feedback Balance Training on Lower Limb Post-Stroke Spasticity, Trunk Performance and Balance:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Emanuela Elena Mihai, Principal Investigator, Carol Davila University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2090/C.E.
Record Dates: First submitted 2021-12-21; First posted 2022-01-19 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic; Spasticity as Sequela of Stroke; Spastic Gait; Balance; Distorted
Keywords: stroke; spasticity; balance trainer; balance impairment; neurologic rehabilitation
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Gait Disorders, Neurologic; Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physiotherapy, visual feedback training, rESWT (Experimental): conventional physiotherapy (5 times/week), visual feedback training (5 times/week), radial extracorporeal shock wave therapy (once/week for 2 weeks)
  Interventions: Other: radial extracorporeal shock wave therapy
- Conventional physiotherapy, visual feedback training, sham rESWT (Sham Comparator): conventional physiotherapy (5 times/week), visual feedback training (5 times/week), sham radial extracorporeal shock wave therapy (once/week for 2 weeks)
  Interventions: Other: sham radial extracorporeal shock wave therapy

INTERVENTIONS:
Other: radial extracorporeal shock wave therapy — rESWT (Endopuls 811; Enraf Nonius B.V. Va-reseweg 127, 3047 AT Rotterdam MedTech, Wessling, Germany) will be applied on the myotendinous junction of both the gastrocnemius and the soleus muscles in post-stroke spasticity patients. 2000 shots will be applied on the gastrocnemius and soleus myotendinous junction with a frequency of 10 Hz and energy density of 60 mJ (1 bar) within tolerable pain limits.
  Arms: Conventional physiotherapy, visual feedback training, rESWT
Other: sham radial extracorporeal shock wave therapy — The control group will receive sound over the myotendinous junction of gastrocnemius and soleus with transducer-like contact.
  Arms: Conventional physiotherapy, visual feedback training, sham rESWT

SUMMARY:
This study assess the relationship between lower limb spasticity and trunk movements during static and dynamic balance in post-stroke patients who also underwent conventional physical therapy, visual feedback balance training and radial extracorporeal shock wave therapy intervention.

DETAILED DESCRIPTION:
The stabilometric assessment through Prokin system complemented the clinical evaluation and provided a more objective, global insight into the combined therapeutic effect.

The stabilometric computerized system is both an assessment tool and a training system for static, dynamic balance and trunk. To date, it was used in various clinical trials as a training tool for promoting stance and balance improvement in several neurorehabilitation programs.

Additional outcomes focused on the effectiveness on pain intensity, clonus, passive range of motion, lower limb sensorimotor function, and functionality. The adverse events were also attentively monitored during the trial.

ELIGIBILITY:
Inclusion Criteria:

* a hemorrhagic or ischemic stroke in acute, subacute or chronic phase;
* no history of previous stroke;
* lower limb post-stroke spasticity and spasticity grade ≥1 on the Modified Ashworth Scale (MAS);
* pain intensity measured on Visual Analogue Scale (VAS) ≥1;
* ability to stand unassisted in upright position for 30 seconds;
* no change in anti-spastic drug dose or treatment and no changes in analgesic medication, as it could affect the results on the Modified Ashworth Scale and the Visual Analogue Scale
* adult patients (>18 years old)

Exclusion Criteria:

* other neurological and orthopaedic disorders or lower limb deformities that could in-terfere with motor performance and balance;
* myopathies;
* severe cognitive impairment, severe aphasia or inability to understand instructions;
* severe spasticity;
* visual field conditions or hemineglect;
* patients unable to undergo follow-up evaluation and excluded from the final analysis;
* anticoagulant medication or any contraindication to receive radial extracorporeal shockwave therapy (rESWT), or any contraindication to physical therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Spasticity grade change | Change from baseline Modified Ashworth Scale at 14 days
  The Modified Ashworth Scale (MAS)

SECONDARY OUTCOMES:
Range of motion change | Change from baseline Passive Range of Motion at 14 days
  passive range of motion (PROM) parameter measured through a hand-held goniometer
Pain intensity change | Change from baseline Visual Analogue Scale at 14 days
  Visual Analogue Scale (VAS) through a vertical 10-cm line (0 - starting pain-free to 10 - the worst imaginable pain). The higher the score means a worse outcome.
Stabilometric outcomes change | Change from baseline Prokin system parameters at 14 days
  Prokin system (PK 252, TecnoBody, Bergamo, Italy) parameters: trunk (degrees), stance (degrees), static (mm^2) and dynamic balance (mm^2)

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Berteanu, Study Director — Physical and Rehabilitation Medicine Department, Elias University Emergency Hospital
Locations (1):
- Elias University Emergency Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No